CLINICAL TRIAL: NCT02107521
Title: The Effect of the Intracytoplasmic Morphologically Selected Sperm Injection in Couples With Previous Implantation Failure After Intracytoplasmic Sperm Injection
Brief Title: IMSI in Couples With Previous Implantation Failures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: broken equipment
Sponsor: Sapientiae Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sapi IMSI IF
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2014-11-18 (Estimated); Status verified 2014-08

CONDITIONS: Male Infertility; Female Infertility
Keywords: sperm morphology; ICSI; IMSI; implantation; pregnancy
MeSH Terms: conditions — Infertility, Male; Infertility, Female | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICSI group (Active Comparator): In this group, sperm selected for injection will be morphologically evaluated under 400x magnification
  Interventions: Other: Intracytoplasmic sperm injection
- IMSI group (Experimental): In this group, sperm selected for injection will be morphologically evaluated under 6600x magnification
  Interventions: Other: Intracytoplasmic morphologically selected sperm injection

INTERVENTIONS:
Other: Intracytoplasmic morphologically selected sperm injection — Sperm selection for injection will be performed at 6600x magnification
  Arms: IMSI group
Other: Intracytoplasmic sperm injection — sperm selection for injection will be performed under 400x magnification
  Arms: ICSI group

SUMMARY:
There is a lack of clarity regarding the justification to instruct the couple to shift from intracytoplasmic sperm injection (ICSI) to intracytoplasmic morphologically selected sperm injection (IMSI). In this study, we aim at evaluating the efficacy of IMSI in couples with previous implantation failure with ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ICSI indication, who have previously underwent >= 1 ICSI attempt in which at least 2 blastocysts were transferred, with no implantation.
* Regular menstrual cycles every 25-35 days.
* Body Mass Index less than 35 as calculated according to the following formula: body weight (kg) / height x height (m2)
* Presence of both ovaries.
* No pelvic and / or clinically significant uterine anomalies.
* Normal cervical cytology.
* Serum follicle stimulating hormone (FSH) within normal limits.

Exclusion Criteria:

* Clinically significant systemic disease.
* Infection by the human immunodeficiency virus (HIV).
* Infection by the by the hepatitis C virus
* Positive test for surface antigens of hepatitis B.
* Endometriosis stages III - IV (classification of the American Society for Reproductive Medicine).
* Hydrosalpinx, unilateral or bilateral.
* Abnormal gynecological bleeding, undiagnosed.
* Allergy or hypersensitivity to human gonadotropin preparations or any other related to the study medication.

-Simultaneous participation in another clinical trial. -

Max Age: 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Implantation | 4-5 weeks' gestation
  The presence of a gestational sac with heart beat, visualized upon ultrasound scan at 4-5 weeks' gestation

CONTACTS AND LOCATIONS:
Overall Officials: Edson Borges, PhD, Principal Investigator — Sapientiae Institute
Locations (1):
- Fertility - Centro de Fertilização Assistida, São Paulo, São Paulo, Brazil